CLINICAL TRIAL: NCT06422117
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase III Study to Evaluate the Efficacy and Safety of HSK16149 Capsule in the Treatment of Moderate to Severe Central Neuropathic Pain in China
Brief Title: Efficacy and Safety of HSK16149 Capsule in the Treatment of Moderate and Severe Central Neuropathic Pain in China
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSK16149-305
Record Dates: First submitted 2024-04-16; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Central Neuropathic Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HSK16149 20mg-40mg bid (Experimental): Oral administration of 20mg twice daily for 12 weeks can be adjusted to 40mg twice daily based on the efficacy and tolerability of the subject
  Interventions: Drug: HSK16149 20mg-40mg BID
- Placebo (Placebo Comparator): Placebo,Oral,2 capsules, twice daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HSK16149 20mg-40mg BID — Oral, 20mg, BID, adjustable to 40mg, BID based on tolerability and efficacy;
  Arms: HSK16149 20mg-40mg bid
Drug: Placebo — Placebo, oral, 2 capsules twice daily
  Arms: Placebo

SUMMARY:
To evaluate the efficacy and safety of HSK16149 capsule in the treatment of moderate to severe central neuropathic pain compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign an informed consent form;
2. Able to read and complete survey questionnaires;
3. Male or female patients aged ≥ 18 years old;
4. The subject has a medical history and symptoms related to central neuropathic pain, including spinal cord related neuropathic pain (subject enrollment ≥ 50%), post-stroke central neuropathic pain, Parkinson's disease pain, and multiple sclerosis pain, and must meet the following criteria: a) pain duration ≥ 3 months; b) Characteristics that conform to neuropathic pain: DN4 scale score ≥ 4 points;
5. During screening visits, patients were assessed to have an average pain visual analogue scale (VAS) score of ≥ 40 mm over the past 24 hours.

Exclusion Criteria:

1. The presence of other painful diseases that may affect the evaluation of neuropathic pain;
2. Patients with spinal cord injury or stroke whose condition is unstable and is expected to require surgical treatment;
3. There is a chronic systemic disease that the investigator has assessed may affect the participant's participation in the study；
4. Meet any of the following laboratory test results: a) Hematology: WBC<3×109/L, N< 1.5 ×109/L, PLT< 75 ×109/L, or HB< 90 g/L; b) Liver function: ALT or AST> 2.5 × ULN; Or TBIL> 1.5 × ULN; c) eGFR< 60 mL/min/1.73 m2; d) Creatine kinase > 2.0 × ULN;
5. Women who are pregnant, planning to become pregnant during the study period, or breastfeeding; Women who do not wish to use reliable contraceptive methods (including condoms, spermicides, or Iuds) for 28 days after signing up for the ICF from the beginning to the last trial drug administration, or who plan to use progesterone contraceptives during this period;
6. Mechanical operators engaged in high-altitude work, motor vehicle driving and other dangerous activities during the study period;
7. Participated in any other clinical study within 30 days prior to screening;
8. The investigator determined that there were other conditions that were not suitable for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Estimated)
Dates: Start 2024-05-30 (Estimated); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-08-07 (Estimated)

PRIMARY OUTCOMES:
The changes of pain scores after treatment in HSK16149 group and placebo group were compared with baseline | week12
  Changes in mean pain intensity (ADPS) at week 12 between HSK16149 and placebo were compared from baseline;The pain NRS score divides a straight line into 10 segments, with 0 to 10 indicating pain (a total of 11 points), 0 indicating no pain, and 10 indicating the most intense pain. The pain NRS scores of the past 7 days were collected and the average value was used as the ADPS score.